CLINICAL TRIAL: NCT06403072
Title: Diagnostic Performance of the Gynecologic Imaging-Reporting and Data System (GI-RADS) in Preoperative Evaluation of Adnexal Masses
Brief Title: (GI-RADS) in Preoperative Evaluation of Adnexal Masses
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Other Study IDs: GI-RADS
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer
Keywords: Gynecologic Imaging-Reporting and Data System; Adnexal Masses; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Gynecologic Imaging-Reporting and Data System (GI-RADS) — The Gynecologic Imaging-Reporting and Data System (GI-RADS) using ultrasound

SUMMARY:
prospective study was conducted and performed on 100 women with pelvic pain due to accidently discovered adnexal mass

DETAILED DESCRIPTION:
After institutional ethical committee approval () and informed consent from the patients, this prospective study was conducted and performed on 100 women with pelvic pain due to accidently discovered adnexal mass

All women were subjected to the following:

1. Detailed history taking: Personal history, Age, Obstetric history, past history and family history.
2. Physical examination: General examination, Pelvic examination and Abdominal examination.
3. Investigations: Routine labs; CBC, liver and kidney functions, FBS and 2HPP. Other labs; cancer antigen 125 (CA 125) as a tumor marker.
4. Trans vaginal ultrasound: TVUS Written informed consent for participation and publication was obtained from each patient after receiving information about the details of the study. Confidentiality of patient's records was assured and maintained throughout the study.

One hundred (100) patients' pelvises were examined by transvaginal ultrasound in lithotomy position using endo-vaginal transducer and/or transabdominal ultrasound in the supine position in transverse and longitudinal plane and evaluated by B-mode ultrasonography, color, and spectral Doppler. Two expert examiners with more than 10 years' experience in gynecological ultrasound, performed all examinations and data was stored between one and four representative images on the database.

After the examinations, a combination of morphological features, color and spectral Doppler features, and then the lesion was evaluated according to GI-RADS classification, and the suggested management protocol based on the risk of malignancy.

Finally, the referral to surgery and decision-making were consulted in accordance with a multidisciplinary team meeting (MDT). A definitive histopathological diagnosis was obtained as a gold standard test for all patients with GI-RADS 4 and 5 and some cases of GI-RADS 3 patients after laparoscopic or surgical removal of the masses.

A morphologic evaluation was performed according to the International Ovarian Tumor Analysis Group (IOTA) recommendations for the following parameters: wall thickness, septation, papillary projections, presence and echogenicity of solid areas, presence of mixed component, cystic component, and presence of ascites and intra-abdominal metastases (peritoneal deposits, liver metastasis, and malignant abdominal lymphadenopathy) was also recorded. Pattern recognition analysis was also used for ovarian masses.

Statistical analysis:

The collected data was coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013 and Microsoft Office Excel 2007.

ELIGIBILITY:
Inclusion Criteria:

* Females complaining of pelvic pain due to adnexal mass

Exclusion Criteria:

* Presence of Sure signs of malignancy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with pelvic pain due to accidently discovered adnexal mass
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The Gynecologic Imaging-Reporting and Data System (GI-RADS) | 1 month from admission to ultrasound investigation and operation and finally histopathology report
  is a reporting system that was created for reporting the findings in adnexal masses based on transvaginal ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Sara S Sara Salem, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided